CLINICAL TRIAL: NCT00941928
Title: Adoptive Transfer of Haploidentical NK Cells in Combination With Epratuzumab for the Treatment of Relapsed Acute Lymphoblastic Leukemia
Brief Title: Haploidentical Natural Killer (NK) Cells With Epratuzumab for Relapsed Acute Lymphoblastic Leukemia (ALL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0160
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Leukemia; Pediatric Cancer
Keywords: Blood And Marrow Transplantation; Relapsed Acute Lymphoblastic Leukemia; ALL; Leukemia; Pediatrics; Haploidentical NK cells; Cyclophosphamide; Cytoxan; Neosar; Epratuzumab; Fludarabine; Fludarabine Phosphate; Fludara; Interleukin-2; IL-2; Proleukin; Low-dose interleukin; Mesna; Mesnex; Natural Killer Cells; NK Cells Transplant
MeSH Terms: conditions — Leukemia; Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — epratuzumab; fludarabine; fludarabine phosphate; Cyclophosphamide; Mesna; Stem Cell Transplantation; IL32 protein, human; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Haploidentical NK cells + Epratuzumab (Experimental): Haploidentical donor-derived NK cell infusion, Epratuzumab 360 mg/m^2 once a day by vein (IV) on Day -4, Day -1 and Days 3, 6, 10, 13 and 17, and low-dose interleukin-2 (IL-2) Subcutaneous injections three times a week for 9 doses on Days 0 to 21; Fludarabine 25 mg/m^2 once a day IV on Day -6 through Day -2 over 30 minutes; Cyclophosphamide 60 mg/kg once a day IV on Days -5 and -4 over 2 hours. Mesna 12 mg/kg by vein 5 times per day on Days -5 and -4 over 15 minutes.
  Interventions: Drug: Epratuzumab; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mesna; Procedure: Infusion of NK cells; Drug: Interleukin-2

INTERVENTIONS:
Drug: Epratuzumab — 360 mg/m^2 once a day by vein on Day -4, Day -1 and Days 3, 6, 10, 13 and 17.
Drug: Fludarabine — 25 mg/m^2 once a day by vein on Day -6 through Day -2 over 30 minutes.
  Other Names: Fludara; Fludarabine Phosphate
Drug: Cyclophosphamide — 60 mg/kg once a day by vein on Days -5 and -4 over 2 hours.
  Other Names: Cytoxan; Neosar
Drug: Mesna — 12 mg/kg by vein 5 times per day on Days -5 and -4 over 15 minutes.
  Other Names: Mesnex
Procedure: Infusion of NK cells — Transplant of Haploidentical NK cells by vein on Day 0.
  Other Names: Stem Cell Transplant; Natural Killer Cells
Drug: Interleukin-2 — Subcutaneous injections three times a week for 9 doses on Days 0 to 21.
  Other Names: IL-2; Proleukin

SUMMARY:
The goal of this clinical research study is to learn if transferring the donor's NK cells, in combination with an antibody called epratuzumab and low-dose interleukin (IL-2), into your body can be done safely. Researchers want to find out if the infused NK cells will survive after the infusion and if the NK cell infusion helps to destroy cancer cells in the recipient's body and possibly to help control the disease.

Primary Objectives:

· Evaluate the feasibility of collecting an adequate number of natural killer (NK) cells from a donor and evaluate the safety of a haploidentical donor-derived NK cell infusion, Epratuzumab, and low-dose interleukin-2 (IL-2).

Secondary Objectives:

* Quantification and persistence of the infused donor NK cell in vivo;
* Quantification and persistence of cytokine levels;
* Assessment of NK cell immunophenotype and function;
* Correlate above with anti-tumor effect.

DETAILED DESCRIPTION:
Study Drugs:

Epratuzumab is designed to attach to certain proteins on the surface of ALL cells. This may cause the cancer cells to die.

Cyclophosphamide is designed to interfere with the multiplication of cancer cells, which may slow or stop their growth. This may cause the cancer cells to die.

Fludarabine is designed to make cancer cells less able to repair damaged DNA (the genetic material of cells). This may increase the likelihood of the cells dying.

IL-2 is designed to help NK cells live longer and work better.

Experimental Therapy:

NK cells are the cells in the body that fight disease and infection. NK cells may destroy tumor cells, particularly when the NK cells are "mismatched" for certain proteins, called human leukocyte antigens (HLA). Researchers think that this ability to destroy tumor cells can be predicted by learning the donor's and the recipient's HLA types to see if they are a mismatch, and by checking for other specialized proteins found on the surface of the donor's NK cells. These proteins are called killer immunoglobulin receptors (KIR).

The NK cells will be collected from the donor's blood and then processed in a lab at M. D. Anderson, where researchers will use a machine, called a CliniMACS device, to separate out the NK cells from the rest of the donor's collected white blood cells and treat them overnight with a drug called IL-2. This is done to make the NK cells stronger before they are given to the recipient. You will also receive IL-2 injections under your skin to try to help the NK cells survive longer and to possibly increase the number of NK cells in your body after the infusion.

Screening Tests:

Before you can start treatment on this study, you will have "screening tests" to help the doctor decide if you are eligible to take part in this study. The following tests and procedures will be performed:

* You will have a bone marrow biopsy and/or aspiration to check the status of the disease. To collect a bone marrow biopsy and/or aspirate, an area of the hip is numbed with an anesthetic, and a small amount of bone marrow and bone is withdrawn through a needle.
* You will have a spinal tap to check the status of the disease. A spinal tap (also called a lumbar puncture) is when a special needle is inserted into the lower back through the space between the bones to draw a sample of the fluid that surrounds the spinal cord.
* You will have a pulse oximetry test to measure your heart rate and the level of oxygen in the blood. To perform this test, a clothespin-shaped device will be placed on your finger for about 1 minute.
* Your medical history will be recorded.
* You will have a physical exam, including a measurement of your vital signs (blood pressure, heart rate, breathing rate, and temperature).
* Blood (about 4 tablespoons) will be drawn for routine tests. This blood will also be checked for infections such as the human immunodeficiency virus (HIV). You will be told the results of this test. If you have an infection, you may not be able to take part in this study.
* Blood (about 2 tablespoons) will be drawn to test for HLA and KIR. You and the donor will be told the results of this test.
* Females who are able to have children must have a negative blood pregnancy test. This test will be performed with the blood drawn for routine tests as described above. If there is not enough blood leftover for this test, additional blood (about 1 teaspoon) will be drawn.

These screening tests, except for the HLA and KIR-typing, would also need to be repeated before an additional leukapheresis procedure can be done as a part of this study, in order to see if you continue to be eligible to have another one performed.

Identifying an Eligible Donor:

Your relative will be tested to see if his or her KIR has a type of "mismatch" that researchers think will help the donor's NK cells target the cancer cells in your body. They must also share half of your HLA genes to be eligible to take part in this study.

The donor's blood will also be checked for infections, such as HIV, to protect against the possibility of transmitting an infection to you during the NK cell infusion.

To help track the NK cells after infusion, researchers prefer (but do not require) that if you are a female recipient, your donor is male and if you are a male recipient, your donor is female.

Epratuzumab Administration:

If you and the donor are found to be eligible to take part in this study, on Day -4 (4 days before the NK cell infusion) and Day -1 (1 day before the NK cell infusion), you will have an epratuzumab infusion. The length of time this infusion will take will be different for each patient. This will be done using an indwelling catheter (a tube that remains in a vein, such as tunneled in the arm or through the chest to continuously inject or drain a part of your body). If you already have an indwelling catheter in place, you will not need to have a new one placed. However, if a new catheter is needed, you will be asked to sign a separate informed consent form for its placement.

On Day -1 (1 day before the NK cell infusion) and on Days 3, 6, 10, 13, and 17, you will receive an epratuzumab infusion. This will take several hours.

Conditioning Phase:

This phase will start within 28 days after the screening tests. During this phase, you will receive chemotherapy with cyclophosphamide and fludarabine to weaken your immune system in order to help the infused NK cells survive. You will stay in the hospital from Day -6 until after the NK cell infusion or longer if the doctor thinks it is necessary.

On Day -6 through Day -2, you will receive fludarabine 1 time each day by vein, over about 30 minutes each time.

On Days -5 and -4, you will receive cyclophosphamide 1 time each day by vein, over about 2 hours each time.

On Days -5 and -4, you will receive mesna 5 times per day by vein, over about 15 minutes each time. Mesna is given to protect your bladder from side effects that may be caused by cyclophosphamide.

Cyclophosphamide, fludarabine, and mesna will all be infused through the same indwelling catheter.

Infusion of NK cells:

On Day 0, you will receive the NK cells by vein, preferably through an indwelling catheter. If you do not have an indwelling catheter, you may receive the infusion intravenously (IV -- by vein). The doctor will decide the amount of NK cells to be infused, which will affect how long the infusion lasts. Usually the infusion should last less than 1 hour.

To help prevent an allergic reaction to the infused NK cells (such as fever and chills), you will receive Benadryl (diphenhydramine) by vein, over 15-30 minutes, and Tylenol (acetaminophen) by mouth. You will also receive fluids by vein to help decrease the risk of kidney damage. If the study doctor thinks it is necessary, you may also receive a steroid to help prevent side effects.

If the doctor thinks that you are not eligible to receive the NK cell infusion on Day 0, you will be taken off study without receiving the donor's NK cells. The collected NK cells will be thrown away.

This study allows eligible recipients under the age of 2 years of age to participate. You and/or a caregiver will be trained how to give the IL-2 injections to yourself. This drug will be injected under the skin for 9 doses. You will take 3 doses per week over a 3-week period after receiving the NK cells.

Measuring NK Cell Survival Through Blood Test:

On Day 0 (before the NK cell infusion and again 2 hours later), and 1 time on each of the following days: Days 2, 7, 14, 21, and 28, blood (about 4 teaspoons each time) will be drawn and tested to see how long the NK cells survive in your body.

If the disease gets worse or the infused NK cells can no longer be seen, this blood draw schedule may be stopped early.

Follow-Up Visits:

You will have follow-up visits at least 3 times per week during the first 3 weeks, and then 1 time about 28 days after your NK cell infusion. Then, you will have additional follow-up visits at about Months 2 and 3. At these visits, the following tests and procedures will be performed:

* You will have any changes in your medical history recorded.
* You will have a physical exam, including a measurement of your vital signs.
* Blood (about 2 tablespoons) will be drawn for routine tests.

On Days 14 and 28, and during Months 2 and 3, you will have a bone marrow biopsy and/or aspiration.

Length of Study:

You will remain on active study for up to 3 months following your NK cell infusion that you agree to have performed.

This is an investigational study. Cyclophosphamide, fludarabine, mesna, and IL-2 are FDA approved and commercially available. Cyclophosphamide and fludarabine are approved for treating leukemia in adults. IL-2 is FDA-approved, but not for the treatment of leukemia.

Epratuzumab is not FDA approved or commercially available. It is only being used in research.

The use of the CliniMACS machine and infusing NK cells combined with epratuzumab in patients with ALL are only being done in research.

Up to 10 recipients and 10 donors will take part in this study. All will be enrolled at The University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Recipient Inclusion criteria (within 28 days of this protocol's lymphodepleting conditioning regimen and after donor and recipient consent-signing)
2. Diagnosis of CD22+ acute lymphoblastic leukemia that is a. refractory to therapy or b. in second or greater relapse without other standard therapeutic options
3. Patient may have been the recipient of an allogeneic hematopoietic stem cell transplant; however; there must be no evidence of Graft-versus-host disease (GVHD)
4. Off prednisone or other immunosuppressive medications for at least 3 days prior to both the lymphodepleting regimen and the NK infusion
5. Zubrod performance scale </= 2 or Lansky performance scale >/= 60
6. Adequate renal function defined as: Serum creatinine (Cr), for adults </= 2 mg/dL, for children </= 2 mg/dL or </= 2 times upper limit of normal (ULN) for age (whichever is less). If abnormal renal function, then Cr clearance >/= 60 mL/min/1.73 m^2
7. Adequate liver function defined as: Total bilirubin </= 2 mg/dL and serum glutamic-pyruvic transaminase (SGPT)/ alanine transaminase(ALT) </= 5 * ULN for age (unless Gilbert's disease or abnormal liver function due to primary disease)
8. Pulmonary symptoms controlled by medication and pulse oximetry >/= 92% room air
9. Negative serum test to rule out pregnancy within 2 weeks prior to registration in females of childbearing potential (non childbearing is defined as greater than one year post-menopausal or surgically sterilized
10. Requirement of sexually active females and males to use any form of contraception considered effective and medically acceptable by the Investigator. [Acceptable forms: birth control implants, birth control pills, a vasectomy (male surgical sterilization), or a double-barrier method (any 2 of the following in combination: intrauterine device (IUD), male or female condom with spermicidal gel, a diaphragm, a sponge, and/or cervical cap)]
11. Negative serology for human immunodeficiency virus (HIV)
12. Donor must be related to recipient and is predicted to be alloreactive based upon the presence of the relevant KIR genes and incompatibility with the recipient for HLA C or Bw antigens
13. Donor must have infectious disease marker testing [Hepatitis B, C, HIV, CMV, Syphilis (RPR), Chagas, HTLV, and West Nile Virus] and CBC differential and platelet studies that meet standard medical eligibility criteria for allogeneic blood stem cell donation within 7 days of apheresis
14. Donor, if a female of childbearing potential (non-childbearing is defined as greater than one year post-menopause or surgically sterilized), must have a negative serum test to rule out pregnancy within 14 days of apheresis
15. Donor must meet standard medical eligibility criteria for allogeneic stem cell donation

Exclusion Criteria:

1. Exclusion criteria applies to both the initiation of conditioning regimen and to the NK infusion
2. Active central nervous system (CNS) leukemia
3. Active infection (defined as on antimicrobial therapy and or febrile)
4. Breast-feeding females
5. Currently using a ventilator or requiring supplemental oxygen
6. Currently undergoing dialysis
7. Currently using a Phase I, II, or III investigational agent. These agents should be stopped within 21 days of NK infusion
8. New detected cardiac arrhythmia not controlled with medical management within prior 72 hour period.
9. Hypotension requiring pressor support within prior 72 hour period
10. Uncontrolled infection defined as daily fever greater than or equal to 38.2°C within prior 24 hours and new positive culture for bacteria, fungus, or virus within 72 hours prior to NK -cell infusion, if clinically indicated
11. Taking corticosteroids by mouth or intravenously within prior 72 hour period
12. Ascites requiring paracentesis within prior 72 hour period. (If the patient requires paracentesis within 72 hours of NK cell infusion, they will not be eligible to receive the infusion.)
13. Seizure activity or clinically detectable encephalopathy or new focal neurologic deficits within prior 72 hour period
14. Donor has active infection (defined as on antimicrobial therapy and/or febrile) within 7 days of apheresis
15. Donor is pregnant female or breast-feeding female (within 7 days of apheresis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Franklin, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 14, 2009 to December 6, 2010. All recruitment occurred at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Haploidentical NK Cells + Epratuzumab: Haploidentical donor-derived NK cell infusion, Epratuzumab 360 mg/m^2 once a day by vein (IV) on Day -4, Day -1 and Days 3, 6, 10, 13 and 17, and low-dose interleukin-2 (IL-2) Subcutaneous injections three times a week for 9 doses on Days 0 to 21; Fludarabine 25 mg/m^2 once a day IV on Day -6 through Day -2 over 30 minutes; Cyclophosphamide 60 mg/kg once a day IV on Days -5 and -4 over 2 hours.
Period: Overall Study
Arm/Group | Haploidentical NK Cells + Epratuzumab
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Haploidentical NK Cells + Epratuzumab
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 11 [6 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: TTP calculated as average time, in months, from baseline to participants disease progression or death, monitored for a minimum of 1 year
Time Frame: 1 Year
Population: Both participants had recurrent disease before single month assessment therefore no data was analyzed. Study was terminated early due to slow accrual.
Arm/Group | Haploidentical NK Cells + Epratuzumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival (OS)
Description: Number of surviving participants without disease progression or death for any reason at one year post treatment.
Time Frame: Minimum of 1 year, or until disease progression or death
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year and 1 month
Arm/Group | Haploidentical NK Cells + Epratuzumab
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical NK Cells + Epratuzumab (N=2)
nausea (General disorders) | 1 (1)
vomitting (Gastrointestinal disorders) | 1 (1)
chills (General disorders) | 1 (1)
pain (Musculoskeletal and connective tissue disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
creatinine phosphokinase increased (Metabolism and nutrition disorders) | 1 (1)
myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
infection (Infections and infestations) | 2 (2)
hypertension (Cardiac disorders) | 1 (1)
cystitis (Renal and urinary disorders) | 1 (1)
hemorrhage, GU (Gastrointestinal disorders) | 1 (1)
muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — muscle weakness of lower limb

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No